CLINICAL TRIAL: NCT05925712
Title: Evaluation of the Clinical Benefits of a Ventilating Suspension Interface for Individuals With Transfemoral Amputation, a Randomized Controlled Cross-over Trial
Brief Title: Aerofit Post Market Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CIP2022020161
Record Dates: First submitted 2023-05-31; First posted 2023-06-29 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Transfemoral Amputation; Amputation; Skin Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Crossover ABA (Experimental): Group 1 starts using the ventilating suspension system (condition A), group 2 starts using non-ventilating suspension system (condition B) and then they cross-over to the other system, two times.
  Interventions: Device: AeroFit Seal-In Liner / Socket; Device: Seal-In Silicone Liner
- Crossover BAB (Experimental): Group 1 starts using the ventilating suspension system (condition A), group 2 starts using non-ventilating suspension system (condition B) and then they cross-over to the other system, two times.
  Interventions: Device: AeroFit Seal-In Liner / Socket; Device: Seal-In Silicone Liner

INTERVENTIONS:
Device: AeroFit Seal-In Liner / Socket — Össur AeroFit® solution is a transfemoral breathable prosthetic interface, combining the AeroFit® Seal-In liner and AeroFit® Socket.
Device: Seal-In Silicone Liner — Seal-In Silicone Lineris transfemoral prosthetic interface used in combination with a prosthetic socket system.

SUMMARY:
The goal of this clinical investigation is to evaluate the clinical benefits of a ventilating suspension interface for individuals with transfemoral amputation. The main aim of the investigation will be to evaluate the clinical user-reported benefits to skin health from using a ventilating lower limb prosthetic suspension system and compare it to a non-ventilating suspension system.

ELIGIBILITY:
Inclusion Criteria:

* 50Kg< body weight < 136Kg
* Cognitive ability to understand all instructions and questionnaires in the study
* Intended for unilateral/bilateral individuals that fit the indications for use, fit within the specified criteria and with the limb length, shape and ability to use a prosthetic liner: Activity level: K1 - K4, Impact level: Low to high, Amputation level: transfemoral
* Congenital transverse deficiency at femoral level
* Using Seal-In Silicone Liner and Direct Socket or AeroFit Seal-In Liner and AeroFit Socket
* Able to use AeroFit Solution, see Figure 7 AeroFit Seal-In Liner Sizes and Figure 8 Minimum socket height per liner profile.
* Residual limb profile: Standard or conical
* Willing and able to participate in the study and follow the protocol
* Confident (all day) prosthetic users for more than 3 months
* Older than 18 years

Exclusion Criteria:

* Participating in another research study that may affect the participation or results of this study (in the opinion of the investigator)
* Users that have received Botox injection as treatment for residual limb sweat issue in the last 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Subject perceived skin health (PEQ-RLH) | 4 weeks
  PEQ-RLH (Prosthesis Evaluation Questionnaire - Residual Limb Health) Questionnaire Mean of six 1-10 point scale items, higher score indicates better RLH

SECONDARY OUTCOMES:
Subject perceived activity restriction and prosthesis use, TAPES-R | 4 weeks
  Self-report: TAPES-R (Trinity Amputation and Prosthesis Experiences Scales) - Activity Restriction scale Mean of ten 3-point scale items, higher score indicates less restriction
Subject perceived quality of life EQ-5D-5L | 4 weeks
  Self-report: EQ-5D-5L 5-level EQ-5D version (EQ-5D-5L) Use of AeroFit system provides non-inferior quality of life* 0-1.00 index value, higher value indicates higher QALY
Incidents of prosthesis slippage, the need to remove liner to dry limb or liner and incidents of complete loss of suspension. | 4 weeks
  Self-report: In-house generated questionnaire on prosthesis slippage and the need to remove prosthesis due to moisture .
  Higher score means worse slippage experience.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Gainesville Prosthetics, Gainesville, Florida
  - NuTech Institute LLC, Indianapolis, Indiana
  - SRT Prosthetics & Orthotics NPC, Indianapolis, Indiana
  - Oakland Orthopedic, Bay City, Michigan
  - Perry Prosthetics, Perrysburg, Ohio
  - Baker Orthotics and Prosthetics, Arlington, Texas
  - Reach Orthotics and Prosthetics Services, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No